CLINICAL TRIAL: NCT02930551
Title: Infiltration of Neuromas With Local Anesthetics to Eliminate Pain: A Double-blinded Crossover Study
Brief Title: Neuromas as the Cause of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Neurom2016
Record Dates: First submitted 2016-09-23; First posted 2016-10-12 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Neuropathic Pain; Neuroma
MeSH Terms: conditions — Neuralgia; Neuroma | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine 2 ml injection with 2% Adrenaline
  Interventions: Drug: Lidocaine
- Isotonic Saline (Placebo Comparator): Isotonic Saline 2 ml Injection
  Interventions: Drug: Isotonic Saline

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine
Drug: Isotonic Saline
  Arms: Isotonic Saline

SUMMARY:
Neuromas are frequent after trauma and surgery, including amputation and can be identified by high-resolution ultrasound. The role of neuromas as the cause of neuropathic pain is uncertain. The investigators therefore wish to explore if spontaneous and evoked pain will be relieved by injection of local anesthetics near painful neuromas in subjects with peripheral nerve injury.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with peripheral nerve injury 3 months prior to participation

Exclusion Criteria:

* Severe somatic or psychiatric diseases
* Other peripheral neuropathy
* Lack of ability to cooperate to the clinical examination
* Allergy to Lidocaine or similar analgetics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Spontaneous pain on numerical rating scale (NRS 0-10) | 15 minutes after injection
  The participant will be asked about spontaneous pain
Evoked pain on numerical rating scale (NRS 0-10) | 15 minutes after injection

SECONDARY OUTCOMES:
Brush allodynia | 15 minutes after injection
  Assesment of area (cm^2) using a SOMEDIC brush
Pinprick hyperalgesia | 15 minutes after injection
  Assesment of area (cm^2) using a von Frey filament (60 g)
Cold allodynia | 15 minutes after injection
  Assesment of area (cm^2) using a roll (20 degrees celcius)
Heat allodynia | 15 minutes after injection
  Assesment of area (cm^2) using a roll (40 degrees celcius)

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No